CLINICAL TRIAL: NCT04306133
Title: Pericapsular Nerve Group (PENG) Block Combined to Wound Infiltration vs. Wound Infiltration Alone for Postoperative Analgesia After Total Hip Replacement: a Prospective Controlled Trial
Brief Title: PENG Block Combined to Wound Infiltration for Hip Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Giuseppe Pascarella, Principal Investigator, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 29/20 PAR ComEt CBM
Record Dates: First submitted 2020-03-08; First posted 2020-03-12 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Postoperative Pain; Analgesia; Hip Arthropathy; Acute Pain; Pain; Postoperative Complications
Keywords: regional anesthesia; hip surgery; PENG
MeSH Terms: conditions — Pain, Postoperative; Agnosia; Acute Pain; Pain; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG BLOCK AND WOUND INFILTRATION (Experimental): Participants receiving PENG block combined to wound infiltration
  Interventions: Procedure: PENG block; Procedure: Wound Infiltration
- WOUND INFILTRATION (Active Comparator): Participants receiving wound infiltration alone
  Interventions: Procedure: Wound Infiltration

INTERVENTIONS:
Procedure: PENG block — After performing spinal anesthesia, PENG block with 20 mL of 0.375 % Ropivacaine will be executed as described by Giron-Arongo et al with a low frequency curvilinear probe. A 22G 80 mm needle (Stimuplex Ultra 360, Braun ) will be used.
  Arms: PENG BLOCK AND WOUND INFILTRATION
Procedure: Wound Infiltration — At the end of operation, the surgeon will perform wound infiltration with 20 mL of 0.375 % Ropivacaine.

SUMMARY:
This study analyze the effect of Pericapsular Nerve Group (PENG) Block combined to wound infiltration for analgesia after elective hip replacement.

Half of participants will receive a PENG Block combined with wound infiltration, while the other half will receive wound infiltration alone.

ELIGIBILITY:
Inclusion Criteria:

* Elective hip replacement surgery
* ASA physical status score < 4

Exclusion Criteria:

* Contraindications to regional anesthesia
* ASA physical status score ≥ 4
* Patient's refusal or inability to sing the informed consent
* Pre-operatively therapy with opioids
* Allergies to any drug provided by the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Maximum Pain Score | 24 hours
  A visual analog pain scale anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]) will be used to evaluate pain during 48 h after surgery
Total opioids consumption | 48 hours
  Total of Sublingual Sufentanil tablets released

SECONDARY OUTCOMES:
Time to first opioid | 48 hours
  Time (hours) from the end of surgery to the first opioid administration
Range of hip motion | 24 hours
  Degrees of hip flexion
Time to ambulation | 48 hours
  Time until the patient is able to stand up and walk with or without assistive devices
Quadriceps weakness | 48 hours
  Presence of weakness of the quadriceps using a scale where 0= no effect; 1 = knee flexion possible but not hip flexion; 2 = absence of knee and hip flexion
Incidence of block complications | 48 hours
  Any complications or side effects of the blocks, such as local infection, intravascular injection of local anesthetics and immediate systemic toxicity.
Opioids side effects | 48 hours
  The presence or absence of opioids side effects such as drowsiness, desaturation, nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Pascarella, MD, Principal Investigator — University Hospital Campus Biomedico of Rome
Locations (1):
- Università Campus Biomedico, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Short AJ, Barnett JJG, Gofeld M, Baig E, Lam K, Agur AMR, Peng PWH. Anatomic Study of Innervation of the Anterior Hip Capsule: Implication for Image-Guided Intervention. Reg Anesth Pain Med. 2018 Feb;43(2):186-192. doi: 10.1097/AAP.0000000000000701. PMID 29140962
- [Result] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Derived] Pascarella G, Costa F, Del Buono R, Pulitano R, Strumia A, Piliego C, De Quattro E, Cataldo R, Agro FE, Carassiti M; collaborators. Impact of the pericapsular nerve group (PENG) block on postoperative analgesia and functional recovery following total hip arthroplasty: a randomised, observer-masked, controlled trial. Anaesthesia. 2021 Nov;76(11):1492-1498. doi: 10.1111/anae.15536. Epub 2021 Jul 1. PMID 34196965